CLINICAL TRIAL: NCT00075452
Title: Phase III Randomized Study Of Gemcitabine Versus Gemcitabine-Oxaliplatine In Patients With Locally Advanced Or Metastatic Pancreatic Carcinoma
Brief Title: Gemcitabine With or Without Oxaliplatin in Treating Patients With Locally Advanced or Metastatic Unresectable Pancreatic Adenocarcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000346480; FRE-GERCOR-GEM-GEMOX/D00-3; EU-20324
Record Dates: First submitted 2004-01-09; First posted 2004-01-12 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2007-05

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage II pancreatic cancer; stage III pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Oxaliplatin

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and oxaliplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether gemcitabine is more effective with or without oxaliplatin in treating pancreatic adenocarcinoma.

PURPOSE: This randomized phase III trial is studying gemcitabine and oxaliplatin to see how well they work compared to gemcitabine alone in treating patients with locally advanced or metastatic unresectable pancreatic adenocarcinoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the overall survival of patients with locally advanced or metastatic unresectable pancreatic adenocarcinoma treated with gemcitabine with or without oxaliplatin.

Secondary

* Compare the time of response in patients treated with these regimens.
* Compare the clinical benefit of and tolerance to these regimens in these patients.
* Compare the quality of life of patients treated with these regimens.
* Compare the progression-free survival of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center, ECOG performance status (0 or 1 vs 2), and extent of disease (locally advanced vs metastatic). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive gemcitabine IV over 30 minutes once weekly on weeks 1-7 and 9-11 in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive gemcitabine IV over 100 minutes on day 1 and oxaliplatin IV over 2 hours on day 2. Courses repeat every 14 days for up to 3 months in the absence of disease progression or unacceptable toxicity.

After the completion of chemotherapy, patients with locally advanced disease receive chemoradiotherapy.

Quality of life is assessed at baseline and then every 2 months.

PROJECTED ACCRUAL: A total of 230 patients (115 per treatment arm) will be accrued for this study within 24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed pancreatic adenocarcinoma

  * Locally advanced or metastatic disease
  * Unresectable disease
* Measurable disease

  * At least 2 cm by a classical scanner and at least 1 cm by a spiral scanner
* No adenocarcinoma of the bile ducts or ampulla of Vater
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 to 75

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* More than 12 weeks

Hematopoietic

* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic

* Bilirubin less than 1.5 times normal
* Alkaline phosphatase less than 5 times normal

Renal

* Creatinine less than 1.5 times normal
* No uncontrolled or persistent hypercalcemia

Cardiovascular

* No serious cardiac failure

Pulmonary

* No serious respiratory failure

Other

* Pain must be stabilized or controlled before initiation of study treatment
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other untreatable malignant tumor
* No serious psychological, familial, social, or geographical condition that would preclude study participation
* No neuropathy that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* No concurrent corticosteroids except for antiemetic therapy

Radiotherapy

* No prior radiotherapy

Surgery

* Not specified

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-11

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Time to response
Clinical benefit
Quality of life
Progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Louvet, MD, PhD — Hopital Saint Antoine
Locations (38):
- France (38):
  - Centre Paul Papin, Angers
  - C.H.G. Beauvais, Beauvais
  - Hopital Saint Andre, Bordeaux
  - CHU Ambroise Pare, Boulogne-Billancourt
  - CMC Bligny, Briis-sous-Forges
  - Hopital Louis Pasteur, Chartres
  - Chu-Hopital Gabriel Montpied, Clermont-Ferrand
  - Hopital Beaujon, Clichy
  - Hopital Louis Mourier, Colombes
  - Hopital Drevon, Dijon
  - Centre Hospitalier Departemental, La Roche-sur-Yon
  - Hopital Saint - Louis, La Rochelle
  - Centre Hospitalier de Lagny, Lagny-sur-Marne
  - Hopital Andre Mignot, Le Chesnay
  - Centre Jean Bernard, Le Mans
  - C. H. Du Mans, Le Mans
  - Hopital Robert Boulin, Libourne
  - Centre Hospital Universitaire Hop Huriez, Lille
  - Clinique Saint Jean, Lyon
  - Hopital de la Croix Rousse, Lyon
  - Hopital Notre-Dame de Bon Secours, Metz
  - Intercommunal Hospital, Montfermeil
  - American Hospital of Paris, Neuilly-sur-Seine
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital Bichat - Claude Bernard, Paris
  - Hopital de la Croix St. Simon, Paris
  - Hopital Saint-Louis, Paris
  - Hopital Saint Antoine, Paris
  - CHU Pitie-Salpetriere, Paris
  - Hopital Tenon, Paris
  - Maison Medicale Marzet, Pau
  - Hopital Haut Leveque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Clinique Ste - Marie, Pontoise
  - Polyclinique De Courlancy, Reims
  - C. H. De Saumur, Saumur
  - C.H. Senlis, Senlis
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Background] Huguet F, Andre T, Hammel P, Artru P, Balosso J, Selle F, Deniaud-Alexandre E, Ruszniewski P, Touboul E, Labianca R, de Gramont A, Louvet C. Impact of chemoradiotherapy after disease control with chemotherapy in locally advanced pancreatic adenocarcinoma in GERCOR phase II and III studies. J Clin Oncol. 2007 Jan 20;25(3):326-31. doi: 10.1200/JCO.2006.07.5663. PMID 17235048
- [Result] Louvet C, Labianca R, Hammel P, Lledo G, Zampino MG, Andre T, Zaniboni A, Ducreux M, Aitini E, Taieb J, Faroux R, Lepere C, de Gramont A; GERCOR; GISCAD. Gemcitabine in combination with oxaliplatin compared with gemcitabine alone in locally advanced or metastatic pancreatic cancer: results of a GERCOR and GISCAD phase III trial. J Clin Oncol. 2005 May 20;23(15):3509-16. doi: 10.1200/JCO.2005.06.023. PMID 15908661